CLINICAL TRIAL: NCT04913272
Title: A Double-Blind, Randomized, Placebo-Controlled Phase 2 Clinical Trial To Evaluate Safety And Efficacy Of KT-301 (Formerly US-APR2020) In Subjects With Chronic Kidney Disease Stage IV
Brief Title: Clinical Trial To Evaluate Safety And Efficacy Of KT-301 (Formerly US-APR2020) In Subjects With Chronic Kidney Disease Stage IV
Acronym: CKD
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistics, company reorganization
Sponsor: Kibow Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: US-APR2020-01
Record Dates: First submitted 2021-05-21; First posted 2021-06-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Kidney Disease stage4

STUDY DESIGN:
Intervention Model Description: This is a Phase 2 double-blind, randomized, placebo-controlled, multicenter clinical trial to evaluate the safety and efficacy of KT-301 (formerly US-APR2020) in patients with CKD Stage IV.
  Following Screening and Enrollment, patients will be Randomized to either Group KT-301 or Placebo. In Group KT-301, the drug KT-301 will be administered orally at 2 capsules per day (one capsule in the morning and one capsule in the evening, after meals, for a total daily dose of 90 Billion CFUs) for six months. Subjects will be followed for 6 months. Patients in Placebo Group will be administered Placebo tablets in similar routine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KT-301 (formerly US-APR2020) (Experimental): Patients in this group will be administered KT-301 (formerly US-APR2020) orally at 2 capsules per day for six months. The frequency will be one capsule in the morning and one capsule in the evening, after meals, (for a total daily dose of 90 Billion CFUs).
  Interventions: Drug: US-APR2020
- Placebo (Placebo Comparator): Patients in this group will be administered placebo orally at 2 capsules per day for six months. The frequency will be one capsule in the morning and one capsule in the evening, after meals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: US-APR2020 — US-APR2020 capsules 45 billion CFUs of the LBT.
  Arms: KT-301 (formerly US-APR2020)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this Phase 2 study is to evaluate the safety and efficacy of the live biotherapeutic product, KT-301 (formerly US-APR2020), in the management of patients with CKD Stage IV.

DETAILED DESCRIPTION:
Kidney diseases are a global public health problem that affects over 200 million people worldwide. It is estimated that about 30 million adults in the United States have Chronic Kidney Disease (CKD) and most are undiagnosed. In addition, CKD represents the ninth leading cause of death in the United States. Kidney diseases also represent great socio-economical cost worldwide. In the United States, treating Medicare beneficiaries with CKD costed over $79 billion, and treating people with End Stage Kidney Disease (ESKD) costed an additional $35 billion in 2016. To date, there is no cure for CKD.

The most important CKD risk factors in adults include diabetes and high blood pressure. Other risk factors include heart disease, obesity, a family history of CKD, past damage to the kidneys, and old age. Having CKD increases the chances of also having heart disease and stroke.

CKD is a condition characterized by a gradual loss of kidney function over time. Depending on the kidney function measured with glomerular filtration rate (GFR) CKD can be classified into several stages (I, II, III, IV and V). CKD Stage V, also known as End Stage Kidney Disease (ESKD), is a very advanced stage of kidney disease where the kidneys have lost nearly all ability to do their job effectively, and eventually dialysis or a kidney transplant is needed to live. Treatment may slow the decline in kidney function and failure. However, not everyone with CKD develops ESKD, and in some cases ESKD develops even with treatment.

CKD is accompanied by altered pathogenic gut bacteria, inflammation, and accumulation of uremic toxins in the blood. These blood uremic toxins can diffuse passively into the bowel. Scientific research has shown that probiotic bacteria could metabolize various uremic toxins such as urea, uric acid, and creatinine. In addition, by supplementing the gut microbiome with probiotic bacteria, it is possible to metabolize the nitrogenous waste products and other toxins which diffuse into the gut, and thus lower levels of inflammation and blood uremic toxins.

KT-301 (formerly US-APR2020) is a live biotherapeutic (LBT) intended to restore the gut microbiome to improve the removal of uremic toxins in the bowel in CKD patients. The aim of this Phase 2 study is to evaluate the safety and efficacy of the KT-301 in the management of patients with CKD Stage IV.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18-80 years
* CKD Stage IV (eGFR = 15-29 mL/min) with declining kidney function for a period > 6 months
* Serum Creatinine > 2.0 mg/dL
* Adherence to low protein diet (LPD) of 0.6-0.8 g/kg/day based on subject response and on advisory

Exclusion Criteria:

* Those on probiotic supplements in the past 3 months
* Pregnancy, breast feeding or females of child-bearing potential who are unwilling to use a reliable form of contraception.
* Immunosuppressant medications therapy specific to immune mediated renal diseases
* HIV/AIDs
* Underweight (BMI ≤ 18.5)
* Subject with an infection that requires oral antibiotic administration at the time of randomization or close to that visit.
* Those with gastrointestinal disease (irritable bowel syndrome or anal fissures or anal fistulas or perianal abscesses or perianal infections or diverticular diseases or colitis or colon polyps) at the time of screening and randomization, or within 6 months prior to the randomization visit (Visit 2)
* Those with internal prosthesis including orthopedics, neurosurgery, heart valves, vascular stents ˂ 2 years post -surgery procedure. Those with Prosthesis > 2 years should not be excluded.
* Those with biological/tissue grafts or prosthesis or implant
* Those on anticoagulant medicines, including Vit K antagonists (e.g., warfarin, coumadin) or the new class of oral anti-coagulants approved by FDA in the last 10 years
* Those on peritoneal dialysis
* Those with acute kidney injury
* Those with mental conditions or medically debilitating disease/disorder other than CKD, which, in the judgment of the investigator, would interfere with or serve as a contraindication to adherence to the study protocol or affect the ability to give informed consent or affect overall prognosis of the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate incidences of Treatment-Emergent Adverse Events following KT-301 (formerly US-APR2020) administration in patients with Chronic Kidney disease (CKD) Stage IV as a measure of safety. | six months
  Presence of adverse events in less than 10% of the study population, as a measure of safety
Evaluate the change of eGFR as per NKF-USFDA guidelines following KT-301 (formerly US-APR2020) administration in patients with Chronic Kidney disease (CKD) Stage IV as a measure of clinical efficacy. | six months
  Arresting the change of Estimated glomerular filtration rate (eGFR) as per National Kidney Foundation- US Food and Drug Administration (NKF-USFDA )guidelines in the group treated with KT-301 (formerly US-APR2020) as compared to the placebo, as a measure of efficacy.

SECONDARY OUTCOMES:
Evaluate changes in basic blood uremic metabolic markers | six months
  Change in any of the basic blood uremic metabolic markers in the group treated with KT-301 (formerly US-APR2020) as compared to the placebo:
  * Blood Urea Nitrogen (BUN)
  * Uric acid
  * Serum creatinine
  * Urea/creatinine ratio
  * Micro albumin urea
Evaluate changes in complete blood count and hematology parameters | six months
  Change in any of the complete blood count (CBC) and hematology parameters in the group treated with KT-301 (formerly US-APR2020) as compared to the placebo:
  * Red blood cells
  * White blood cells
  * Platelets
  * Hemoglobin (Hgb)
  * Hematocrit (Hct) Ferritin
Evaluate changes in C-Reactive Protein (CRP) levels | six months
  Change in C-Reactive Protein (CRP) levels in the group treated with KT-301 (formerly US-APR2020) as compared to the placebo
Evaluate change in quality of life (QOL)- SF36 QOL questionnaire | six months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Jadedstone Clinical Research, Silver Spring, Maryland
  - Kidney Michigan, Saginaw, Michigan
  - South Carolina Clinical Research, Orangeburg, South Carolina
  - Almeda Medical Clinic, Houston, Texas
  - Mendez Center for Clinical Research, Woodbridge, Virginia